CLINICAL TRIAL: NCT05128279
Title: Analysis of Corrections of Adolescent and Young Adulte Scoliosis by Posterior Instrumentation
Brief Title: Adolescent and Young Adulte Scoliosis
Acronym: AIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7961
Record Dates: First submitted 2021-10-20; First posted 2021-11-19 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; Thoracic hyperkyphosis; Cyphosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thoracic hypocyphosis and greater lumbar lordosis after correction of idiopathic scoliosis in adolescents and young adults may adversely affect overall sagittal alignment and increase the risk of proximal junctional kyphosis.

The objective of this study is to analyze surgical corrections and maintenance of correction over time using modern posterior instrumentation strategies by comparing technical developments.

ELIGIBILITY:
Inclusion criteria:

* Major subjects> 18 years old
* Subject with a surgical indication for arthrodesis and surgical correction of adolescent or young adult scoliosis
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subjects with a surgical indication for arthrodesis and surgical correction of adolescent or young adult scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03-18 (Estimated)

PRIMARY OUTCOMES:
Study of corrections of adolescent and young adult scoliosis by posterior instrumentation | Files analysed retrospectively from January 01, 2010 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie du Rachis - Hôpitaux Universitaires de Strasbourg, Strasbourg, France